CLINICAL TRIAL: NCT02920255
Title: Comparison of Electronic Caliper Measurements of Spinal Tilt to Conventional Caliper and X-ray Measurements of Spinal Tilt
Brief Title: Comparison of Electronic Calipers to Conventional Calipers and X-ray Measurement of Spinal Tilt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KKT Orthopedic Spine Center (Industry)
Responsible Party: Sponsor
Other Study IDs: Caliper 1001
Record Dates: First submitted 2016-09-22; First posted 2016-09-30 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Electronic Caliper Measurements: This arm would be the spinal diagnostic measurements taken at the hips and shoulders of participants with electronic calipers.
  Interventions: Other: Diagnostic
- Conventional Caliper Measurements: This arm would be the spinal diagnostic measurements taken at the hips and shoulders of participants with conventional calipers.
  Interventions: Other: Diagnostic
- X-ray Measurements: This arm would be the spinal diagnostic measurements taken at the hips and shoulders of participants with x-rays.
  Interventions: Other: Diagnostic

INTERVENTIONS:
Other: Diagnostic — Measurement of spinal tilt

SUMMARY:
The objective is to compare the accuracy and reproducibility of measurements taken with electronic calipers and conventional calipers. Using both calipers, reproducibility will be determined by comparing results from a number of practitioners and accuracy will be determined by comparing results with those obtained from X-rays.

DETAILED DESCRIPTION:
Participants will have 2 spinal measurements, one at the shoulder and one at the hip, taken by electronic calipers and conventional calipers with different individual research staff. Up to 5 individual research staff will take the 2 spinal measurements on each participant. This will be done to compare variation of measurements between individual operators.

The accuracy of the spinal measurements, obtained with electronic and conventional calipers will be compared to the results obtained from x-rays taken of shoulder and hip areas. Only one x-ray of the shoulder and one x-ray of the hip will be taken of each participant. X-rays represent the clinically accepted standard of obtaining spinal measurements.

The data will analyzed statistically to determine sources of variation among the methods of spinal measurement described above.

ELIGIBILITY:
Inclusion Criteria

Must be able to have shoulder and hip measurements for spinal tilt

Exclusion Criteria:

Not able to have shoulder and and hip measurements for spinal tilt.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient Population and Normal Volunteers at KKT Orthopedic Spinal Center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Electronic Caliper Spinal Measurements | Through study completion, an average of 13 months
  All measurements will recorded in degrees of spinal tilt.

SECONDARY OUTCOMES:
Accuracy of Conventional Caliper Spinal Measurements | Through study completion, an average of 13 months
  All measurements will recorded in degrees of spinal tilt.
Accuracy of X-ray Spinal Measurements | Through study completion, an average of 13 months
  All measurements will recorded in degrees of spinal tilt.
Reproducibility of Electronic Caliper Measurements | Through study completion, an average of 13 months
  All measurements will recorded in degrees of spinal tilt.
Reproducibility of Conventional Caliper Measurements | Through study completion, an average of 13 months
  All measurements will recorded in degrees of spinal tilt.
Reproducibility of X-ray Measurements | Through study completion, an average of 13 months
  All measurements will recorded in degrees of spinal tilt.

CONTACTS AND LOCATIONS:
Overall Officials: Aslam Khan, DC, Principal Investigator — KKT Orthopedic Spine Center
Locations (1):
- KKT Orthopedic Spine Center, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akel I, Pekmezci M, Hayran M, Genc Y, Kocak O, Derman O, Erdogan I, Yazici M. Evaluation of shoulder balance in the normal adolescent population and its correlation with radiological parameters. Eur Spine J. 2008 Mar;17(3):348-354. doi: 10.1007/s00586-007-0546-0. Epub 2007 Nov 20. PMID 18027001